CLINICAL TRIAL: NCT02978196
Title: 99mTc/68Ga Labeled Anti-PD-L1 sdAb in Assessment of Programmed Death Ligand-1 Expression in Non-small Cell Lung Cancer
Brief Title: 99mTc/68Ga Labeled Anti-PD-L1 sdAb in Assessment of PD-L1 Expression in NSCLC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: NanoMab Technology (UK) Limited (Industry)
Responsible Party: Principal Investigator, Zhao Jin Hua, MD, Director Department of Nuclear Medicine, Principal Investigator, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: [2019]310
Record Dates: First submitted 2016-11-22; First posted 2016-11-30 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injection of 99mTc-NM-01 (Experimental): All patients with NSCLC who have undergone biopsy of primary tumour lesion will be administered 3-12 MBq/kg of 99mTc-NM-01 in a single injection.
  Interventions: Procedure: Injection of 99mTc-NM-01
- Injection of 68Ga-NM-01 (Experimental): All patients with NSCLC who have undergone biopsy of primary tumour lesion will be administered 0.75- 4 MBq/kg of 68Ga-NM-01 in a single injection.
  Interventions: Procedure: Injection of 68Ga-NM-01

INTERVENTIONS:
Procedure: Injection of 99mTc-NM-01 — Patient is injected with micro-dose of 99mTc-NM-01
  Arms: Injection of 99mTc-NM-01
Procedure: Injection of 68Ga-NM-01 — Patient is injected with micro-dose of 68Ga-NM-01
  Arms: Injection of 68Ga-NM-01

SUMMARY:
To evaluate the safety, dosimetry and efficacy of 99mTc/68Ga labeled anti-PD-L1 single domian antibody (sdAb) (Product Code Name: 99mTc-NM-01 and 68Ga-NM-01) in the diagnostic imaging PD-L1 expression in Non-Small Cell Lung Cancer (NSCLC) and compare it with the existing gold standard "biopsy PD-L1 detection". It is also to establish a new clinical method of non-invasive PD-L1 expression detection in NSCLC using 99mTc/68Ga labeled anti-PD-L1 sdAb.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for the participation in the study before any protocol-specific screening procedures are performed
* Male or female, aged 18-75 years old
* Previous diagnosis of non-small cell carcinoma, confirmed with pathology tests
* AST, ALT, BUN, Cr not more than double the normal values
* Patients with no current history of hepatitis A, hepatitis B, AIDS, tuberculosis and other infectious diseases

Exclusion Criteria:

* Severe infection
* Unable to provide biopsy sample for testing PD-L1 expression level
* Patients with pacemakers
* Pregnant and lactating women
* Investigators professional decision that the subject should not participate in this clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Assessment of PD-L1 expression in NSCLC using 99mTc-NM-01 SPECT/CT and 68Ga-NM-01 PET/CT Scan | 1 year
  Visual analysis will be carried out by 4 experienced nuclear medicine physicians to observe the uptake of 99mTc-NM-01 and 68Ga-NM-01 in lung lesions. A 4 point system will be used to interpret the scans for abnormalities. It is categorised as such: score 0, no abnormal increased uptake; score 1, low increased uptake; score 2, moderate increased uptake; score 3, high increased uptake. The lesion will be considered positive for malignancy if the score is 2 or higher.
Semiquantitative Assessment of Lung Lesions in 99mTc-NM-01 SPECT/CT and 68Ga-NM-01 PET Scan | 1 year
  Patients in the 99mTc-NM-01 group will be administered 3-12 MBq/kg of 99mTc-NM-01 and patients in the 68Ga-NM-01 group will be administered 0.75-4 MBq/kg of 68Ga-NM-01. The semiquantitative analysis of the region of interest (ROI) will be performed in lung lesions. Higher level of PD-L1 expression (Tumor proportion score, TPS), higher ROI in tumor. No expression TPS < 1%; Low expression TPS 1 - 49%; High expression TPS ≥ 50%.

SECONDARY OUTCOMES:
PD-L1 expression levels | 1 year
  Patients biopsy sample will be tested to confirm the levels of PD-L1 expression using Human PD-L1 ELISA Kit.
Adverse Drug Reaction Report | 7 days
  Monitor adverse events within 7 days after the injection and scanning to establish the safety of 99mTc-NM-01 and 68Ga-NM-01 in patients.
New tumor lesion detection | 1 year
  99mTc-NM-01 SPECT/CT and 68Ga-NM-01 PET/CT may detect new tumor areas, which can be further proven by biopsy method in order to rule out any false positive results.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, China

REFERENCES:
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Brahmer JR, Drake CG, Wollner I, Powderly JD, Picus J, Sharfman WH, Stankevich E, Pons A, Salay TM, McMiller TL, Gilson MM, Wang C, Selby M, Taube JM, Anders R, Chen L, Korman AJ, Pardoll DM, Lowy I, Topalian SL. Phase I study of single-agent anti-programmed death-1 (MDX-1106) in refractory solid tumors: safety, clinical activity, pharmacodynamics, and immunologic correlates. J Clin Oncol. 2010 Jul 1;28(19):3167-75. doi: 10.1200/JCO.2009.26.7609. Epub 2010 Jun 1. PMID 20516446
- [Background] Zhang J, Gao J, Li Y, Nie J, Dai L, Hu W, Chen X, Han J, Ma X, Tian G, Wu D, Shen L, Fang J. Circulating PD-L1 in NSCLC patients and the correlation between the level of PD-L1 expression and the clinical characteristics. Thorac Cancer. 2015 Jul;6(4):534-8. doi: 10.1111/1759-7714.12247. Epub 2015 Mar 5. PMID 26273411
- [Background] Heskamp S, Hobo W, Molkenboer-Kuenen JD, Olive D, Oyen WJ, Dolstra H, Boerman OC. Noninvasive Imaging of Tumor PD-L1 Expression Using Radiolabeled Anti-PD-L1 Antibodies. Cancer Res. 2015 Jul 15;75(14):2928-36. doi: 10.1158/0008-5472.CAN-14-3477. Epub 2015 May 14. PMID 25977331
- [Background] Josefsson A, Nedrow JR, Park S, Banerjee SR, Rittenbach A, Jammes F, Tsui B, Sgouros G. Imaging, Biodistribution, and Dosimetry of Radionuclide-Labeled PD-L1 Antibody in an Immunocompetent Mouse Model of Breast Cancer. Cancer Res. 2016 Jan 15;76(2):472-9. doi: 10.1158/0008-5472.CAN-15-2141. Epub 2015 Nov 10. PMID 26554829
- [Derived] Zhao L, Gong J, Liao S, Huang W, Zhao J, Xing Y. Preclinical evaluation and preliminary clinical study of 68Ga-NODAGA-NM-01 for PET imaging of PD-L1 expression. Cancer Imaging. 2025 Jan 27;25(1):6. doi: 10.1186/s40644-025-00826-8. PMID 39871394
- [Derived] Hughes DJ, Chand G, Goh V, Cook GJR. Inter- and intraobserver agreement of the quantitative assessment of [99mTc]-labelled anti-programmed death-ligand 1 (PD-L1) SPECT/CT in non-small cell lung cancer. EJNMMI Res. 2020 Dec 1;10(1):145. doi: 10.1186/s13550-020-00734-x. PMID 33259032 (Retraction: PMID 34637006 EJNMMI Res. 2021 Oct 12;11(1):102)